CLINICAL TRIAL: NCT04856501
Title: A Randomized Control Trial of a Responsive Parenting Intervention to Support Healthy Brain Development and Self-regulation in Toddlers Born Preterm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Herman H. Fleishman Foundation (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Dana DeMaster, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-17-0190; 1R01HD100560-01A1 (NIH)
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PALS intervention condition (Experimental)
  Interventions: Behavioral: PALS intervention condition
- Control condition (Active Comparator)
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: PALS intervention condition — The Play and Learning Strategies (PALS) intervention provides parents with behaviors that, collectively, are known as a responsive parenting style. Four constructs make up this responsive parenting style: 1) contingent responsiveness, (responses are conditionally linked to the child's signals) 2) warm sensitivity (high levels of affection and understanding of child states), 3) maintaining vs. redirecting attention, and 4) verbal scaffolding (providing child appropriate language supports). Parents assigned to this intervention will be paired with a coach who will guide them through the program over the course of 9 weekly sessions. The intervention (ePALS) will be implemented via an internet adaptation through the Children's Learning Institute's ENGAGE platform. However, ePALS could easily be adapted for other platforms and accessed with any web-enabled device.
  Arms: PALS intervention condition
Behavioral: Control condition — Families assigned to the control condition will be provided with a website with information corresponding to milestones of toddler development. Control families will be asked to review that week's materials before the each of the 9 weekly coach calls. The active control condition serves three important purposes: 1) Maintains an active line of communication and accurate contact records for Post-test 1 and Post-test 2 session scheduling; 2) Masks participant's awareness of intervention vs. control assignment; and 3) Approximates communication with intervention staff such that results showing ePALS effects are attributable to intervention rather than regular communication with an interventionist.
  Arms: Control condition

SUMMARY:
The purpose of this study is to determine whether participation in the Play and Learning Strategies (PALS) parenting intervention results in increased caregiver responsiveness behaviors and to test if participation in PALS results in increases in toddler skills and/or toddler neurological development.

ELIGIBILITY:
Inclusion Criteria:

- Maternal age over 18-years when child was born

Exclusion Criteria:

* presence of known/suspected congenital anomalies including chromosomal or complex congenital heart disease
* congenital infection including TORCH (Toxoplasmosis, Rubella, Cytomegalovirus, Herpes Simplex and others),untreated maternal HIV, or maternal syphilis
* bilateral grade 3/4 intraventricular hemorrhage,intraparenchymal hemorrhage, hydrocephalus
* Cerebral palsy with Gross Motor Function Classification of III or higher
* blindness-
* deafness
* Current maternal drug use or maternal drug use during pregnancy
* families who reside outside the catchment area (>1 hour drive from the Texas Medical Center)
* Child with contraindication for MRI. If the mother of the child is pregnant, thinks she might be pregnant, or has a contraindication for MRI, another relative of the child will be asked to assist with the MRIs

Ages: 15 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Parental contingent responsiveness as measured by the Parent-child Toy Play Observation | Baseline, Post-test 1 (1-2 weeks after intervention)
  In this task the child will interact with their parent in a "free play" task for 10 minutes with a set of standardized toys, and the interaction will be videotaped. Parents are asked to play with their children in "typical ways" with a few constraints (e.g., television must be off). Behavior will be coded and assigned a score of how of 1-5 which indicates how often the assessed behavior occurs: 5 (Almost Always); 4 (greater than half the time); 3 (half the time); 2 (less than half the time); 1 (None of the time).
Change in Parental warm sensitivity (display of positive affect) as measured by the Parent-child Toy Play Observation | Baseline, Post-test 1 (1-2 weeks after intervention)
  In this task the child will interact with their parent in a "free play" task for 10 minutes with a set of standardized toys, and the interaction will be videotaped. Parents are asked to play with their children in "typical ways" with a few constraints (e.g., television must be off). Behavior will be coded and assigned a score of how of 1-5 which indicates how often the assessed behavior occurs: 5 (Almost Always); 4 (greater than half the time); 3 (half the time); 2 (less than half the time); 1 (None of the time).
Change in Parental warm sensitivity (warmth) as measured by the Parent-child Toy Play Observation | Baseline, Post-test 1 (1-2 weeks after intervention)
  In this task the child will interact with their parent in a "free play" task for 10 minutes with a set of standardized toys, and the interaction will be videotaped. Parents are asked to play with their children in "typical ways" with a few constraints (e.g., television must be off). Behavior will be coded and assigned a score of how of 1-5 which indicates how often the assessed behavior occurs: 5 (Almost Always); 4 (greater than half the time); 3 (half the time); 2 (less than half the time); 1 (None of the time).
Change in Parental maintaining of child's signals and interests as measured by the Parent-child Toy Play Observation | Baseline, Post-test 1 (1-2 weeks after intervention)
  In this task the child will interact with their parent in a "free play" task for 10 minutes with a set of standardized toys, and the interaction will be videotaped. Parents are asked to play with their children in "typical ways" with a few constraints (e.g., television must be off). Behavior will be coded and assigned a score of how of 1-5 which indicates how often the assessed behavior occurs: 5 (Almost Always); 4 (greater than half the time); 3 (half the time); 2 (less than half the time); 1 (None of the time).
Change in Parental verbal scaffolding as measured by the Parent-child Toy Play Observation | Baseline, Post-test 1 (1-2 weeks after intervention)
  In this task the child will interact with their parent in a "free play" task for 10 minutes with a set of standardized toys, and the interaction will be videotaped. Parents are asked to play with their children in "typical ways" with a few constraints (e.g., television must be off). Behavior will be coded and assigned a score of how of 1-5 which indicates how often the assessed behavior occurs: 5 (Almost Always); 4 (greater than half the time); 3 (half the time); 2 (less than half the time); 1 (None of the time).
Change in Child attentional engagement (engagement with environment) as measured by the Parent-child Toy Play Observation | Baseline, Post-test 1 (1-2 weeks after intervention)
  In this task the child will interact with their parent in a "free play" task for 10 minutes with a set of standardized toys, and the interaction will be videotaped. Parents are asked to play with their children in "typical ways" with a few constraints (e.g., television must be off). Behavior will be coded and assigned a score of how of 1-5 which indicates how often the assessed behavior occurs: 5 (Almost Always); 4 (greater than half the time); 3 (half the time); 2 (less than half the time); 1 (None of the time).
Change in Child attentional engagement (social engagement) as measured by the Parent-child Toy Play Observation | Baseline, Post-test 1 (1-2 weeks after intervention)
  In this task the child will interact with their parent in a "free play" task for 10 minutes with a set of standardized toys, and the interaction will be videotaped. Parents are asked to play with their children in "typical ways" with a few constraints (e.g., television must be off). Behavior will be coded and assigned a score of how of 1-5 which indicates how often the assessed behavior occurs: 5 (Almost Always); 4 (greater than half the time); 3 (half the time); 2 (less than half the time); 1 (None of the time).
Change in Child emotional regulation as measured by the Parent-child Toy Play Observation | Baseline, Post-test 1 (1-2 weeks after intervention)
  In this task the child will interact with their parent in a "free play" task for 10 minutes with a set of standardized toys, and the interaction will be videotaped. Parents are asked to play with their children in "typical ways" with a few constraints (e.g., television must be off). Behavior will be coded and assigned a score of how of 1-5 which indicates how often the assessed behavior occurs: 5 (Almost Always); 4 (greater than half the time); 3 (half the time); 2 (less than half the time); 1 (None of the time).
Change in Child cooperation as measured by the Parent-child Toy Play Observation | Baseline, Post-test 1 (1-2 weeks after intervention)
  In this task the child will interact with their parent in a "free play" task for 10 minutes with a set of standardized toys, and the interaction will be videotaped. Parents are asked to play with their children in "typical ways" with a few constraints (e.g., television must be off). Behavior will be coded and assigned a score of how of 1-5 which indicates how often the assessed behavior occurs: 5 (Almost Always); 4 (greater than half the time); 3 (half the time); 2 (less than half the time); 1 (None of the time).
Change in Child emotional regulation (proximity seeking behaviors) as assessed by score on Waiting Task | Baseline, Post-test 1 (1-2 weeks after intervention)
  This task measures child frustration and parenting behaviors related to child's frustration. During this assessment the assessor provides the parent paperwork to complete and places an elaborately wrapped gift on the table in front of the child. The parent is instructed to have the child wait to open the gift until the assessor returns to the room and then the parent and child are left alone in a room for 8 minutes. Behavior is coded and scored.A score of 1 to 5 will be assigned to indicate how often the behavior occurred, as follows: 1 = 0 reaches; 2 = 1 - 2 reaches that are 15sec. sustained; 3 = 3 reaches that are 30sec. sustained; 4 = 4 Individually scored reaches that are 45sec. sustained; 5 = 5 or more reaches that are 60sec.
Change in Child emotional regulation (venting/aggression/distress behaviors) as assessed by score on Waiting Task | Baseline, Post-test 1 (1-2 weeks after intervention)
  This task measures child frustration and parenting behaviors related to child's frustration. During this assessment the assessor provides the parent paperwork to complete and places an elaborately wrapped gift on the table in front of the child. The parent is instructed to have the child wait to open the gift until the assessor returns to the room and then the parent and child are left alone in a room for 8 minutes. Behavior is coded and scored. A score of 1 to 5 will be assigned to indicate how often the behavior occurred, as follows: 1 = did not happen; 2 = 1 brief instance -15 sec. sustained; 3 = 2 - 3 times -30 sec. sustained; 4 = ¾ instances - 45 sec. sustained; 5 = spends most of minute - >45 sec.
Change in Child emotional regulation (disengaged behavior) as assessed by score on Waiting Task | Baseline, Post-test 1 (1-2 weeks after intervention)
  This task measures child frustration and parenting behaviors related to child's frustration. During this assessment the assessor provides the parent paperwork to complete and places an elaborately wrapped gift on the table in front of the child. The parent is instructed to have the child wait to open the gift until the assessor returns to the room and then the parent and child are left alone in a room for 8 minutes. Behavior is coded and scored. A score of 1 to 5 will be assigned to indicate how often the behavior occurred, as follows: 1 = 0 sec.; 2 = 15 sec. sustained; 3 = 30 sec sustained; 4 = 45 sec sustained; 5 = 60 sec sustained
Change in Child inhibition (verbal distraction) as assessed by score on Waiting Task | Baseline, Post-test 1 (1-2 weeks after intervention)
  This task measures child frustration and parenting behaviors related to child's frustration. During this assessment the assessor provides the parent paperwork to complete and places an elaborately wrapped gift on the table in front of the child. The parent is instructed to have the child wait to open the gift until the assessor returns to the room and then the parent and child are left alone in a room for 8 minutes. Behavior is coded and scored.A score of 1 to 5 will be assigned to indicate how often the behavior occurred, as follows: 1 = did not happen; 2 = 1 brief instance; 3 = 2/3 times w/ sustaining behavior; 4 = 3/4 times w/ sustained behavior; 5 = spends most of minute trying to get parent attention in appropriate way
Change in Child inhibition (self-distraction) as assessed by score on Waiting Task | Baseline, Post-test 1 (1-2 weeks after intervention)
  This task measures child frustration and parenting behaviors related to child's frustration. During this assessment the assessor provides the parent paperwork to complete and places an elaborately wrapped gift on the table in front of the child. The parent is instructed to have the child wait to open the gift until the assessor returns to the room and then the parent and child are left alone in a room for 8 minutes.Behavior is coded and scored A score of 1 to 5 will be assigned to indicate how often the behavior occurred, as follows: 1 = did not happen; 2 = 1 occurrence; 3 = 2/3 occurrences; 4 = 4 occurrences; 5 = 5 or more occurrences
Change in number of times parent exhibit warm sensitivity (physical soothing behaviors) as measured by the Waiting Task | Baseline, Post-test 1 (1-2 weeks after intervention)
  This task measures child frustration and parenting behaviors related to child's frustration. During this assessment the assessor provides the parent paperwork to complete and places an elaborately wrapped gift on the table in front of the child. The parent is instructed to have the child wait to open the gift until the assessor returns to the room and then the parent and child are left alone in a room for 8 minutes. Number of times parent exhibits the behavior will be reported.
Change in number of times parent exhibits parental verbal scaffolding (verbal distraction behaviors) as measured by the Waiting Task | Baseline, Post-test 1 (1-2 weeks after intervention)
  This task measures child frustration and parenting behaviors related to child's frustration. During this assessment the assessor provides the parent paperwork to complete and places an elaborately wrapped gift on the table in front of the child. The parent is instructed to have the child wait to open the gift until the assessor returns to the room and then the parent and child are left alone in a room for 8 minutes. Number of times parent exhibits the behavior will be reported.
Change in number of times parent exhibits parental contingent responsiveness (responsive behavior - promotion behaviors) as measured by the Waiting Task | Baseline, Post-test 1 (1-2 weeks after intervention)
  This task measures child frustration and parenting behaviors related to child's frustration. During this assessment the assessor provides the parent paperwork to complete and places an elaborately wrapped gift on the table in front of the child. The parent is instructed to have the child wait to open the gift until the assessor returns to the room and then the parent and child are left alone in a room for 8 minutes. Number of times parent exhibits the behavior will be reported.
Change in Number of times parent exhibits non-responsive behavior(prevention behaviors) as measured by the Waiting Task | Baseline, Post-test 1 (1-2 weeks after intervention)
  This task measures child frustration and parenting behaviors related to child's frustration. During this assessment the assessor provides the parent paperwork to complete and places an elaborately wrapped gift on the table in front of the child. The parent is instructed to have the child wait to open the gift until the assessor returns to the room and then the parent and child are left alone in a room for 8 minutes. Number of times parent exhibits the behavior will be reported.
Change in number of times parent exhibits parental non-responsive behavior(destructive coping and harsh physical restraint behaviors) as measured by the Waiting Task | Baseline, Post-test 1 (1-2 weeks after intervention)
  This task measures child frustration and parenting behaviors related to child's frustration. During this assessment the assessor provides the parent paperwork to complete and places an elaborately wrapped gift on the table in front of the child. The parent is instructed to have the child wait to open the gift until the assessor returns to the room and then the parent and child are left alone in a room for 8 minutes. Number of times parent exhibits the behavior will be reported.
Change in Childs problem solving skill as measured by the Independent Toy Play task | Baseline, Post-test-2 (4 months after post test1)
  This task measures child skill related to problem solving through goal-directed play. For this task, the child is videotaped while playing alone with five sequentially presented toys, each presented for 2mins. The video will be subsequently coded by dividing the play session into 10 second intervals. Level of the child's play is coded based on a hierarchical level-of-play scale ranging from 1 (off task) to 13 (goal-directed play with mastery).
Change in Child working memory as assessed by the 3-6-9 box task | Baseline, Post-test-2 (4 months after post test1)
  This task measures child working memory. During the task, children are asked to search 3-, then 6-, then 9- box arrays for hidden rewards. Children are asked to search individual boxes in the array one at a time and to keep track of the boxes that were previously searched. Between each search attempt, the boxes are covered which requires children to remember which boxes were previously searched. The task begins with a 3-box array where children are given 10 trials to find three rewards. Children who complete the 3-box array will move on to a 6-box array where they will have 20 trials to locate six rewards. Children will only progress to the nine-box array (max. 30 trials) if the six-box array is completed in 14 trials or less. Score is reported as the number of rewards found divided by the number of total reaches.
Change in Child's self-restraint as assessed by score on the Gift Wrap step of the Gift Wrap/Waiting for Bow task | Baseline, Post-test-2 (4 months after post test1)
  In this assessment, children are seated across a table from an assessor and are told that they will receive a present but that the present must be wrapped. The experimenter asks that the child turns their back and does not peek while she wraps the present because seeing it ruins the surprise. While the child is turned away, the experimenter noisily wraps for 1 minute. After this portion is complete, the experimenter tells the child that she forgot to put a bow on the gift, and asks the child to wait and not touch the box until she returns with a bow. The experimenter leaves for 2 minutes. Child's self-restraint is scored from 0-3 where 0 = no peeking, 1=Child looks over shoulder to peek, 2=child turns body in seat to peek, and 3 = child left her seat.
Change in Child's self-restraint as assessed by score on the Waiting for Bow step of the Gift Wrap/Waiting for Bow task | Baseline, Post-test-2 (4 months after post test1)
  In this assessment, children are seated across a table from an assessor and are told that they will receive a present but that the present must be wrapped. The experimenter asks that the child turns their back and does not peek while she wraps the present because seeing it ruins the surprise. While the child is turned away, the experimenter noisily wraps for 1 minute. After this portion is complete, the experimenter tells the child that she forgot to put a bow on the gift, and asks the child to wait and not touch the box until she returns with a bow. The experimenter leaves for 2 minutes. Child's self-restraint is scored from 0-4 where 0 = no touching, 1 = child touches box, 2 = Child opens the box so that the lid is less than 2 inches from base; looks and then replaces lid, 3 = Child opens the box or child completely removes lid from box, and 4 = child removes the toy from the box or child touches the toy while it remains in the box.
Change in Child's distraction as assessed by score in the Waiting for Bow step of the Gift Wrap/Waiting for Bow task | Baseline, Post-test-2 (4 months after post test1)
  In this assessment, children are seated across a table from an assessor and are told that they will receive a present but that the present must be wrapped. The experimenter asks that the child turns their back and does not peek while she wraps the present because seeing it ruins the surprise. While the child is turned away, the experimenter noisily wraps for 1 minute. After this portion is complete, the experimenter tells the child that she forgot to put a bow on the gift, and asks the child to wait and not touch the box until she returns with a bow. The experimenter leaves for 2 minutes. Child's distraction is scored from 0-5 where 1 = no active actions, 2 = a little bit of time, 3 = Some of the time, 4 = a lot of the time, 5 = most of the time.
Change in Noncompliance behaviors of child toward parent as measured by the Tool task | Baseline, Post-test-2 (4 months after post test1)
  The parent and child complete two problem solving tasks that are graded in difficulty. The assessor explains the problem to the parent and gives the tool and apparatus to the child. The parent is instructed to allow the child to solve the problem independently, but provide as much help as they believe the child needs. Task 1 is the "tube task", in which the child has to insert a stick inside a tube to get a toy. Task 2 is the "clear box task" that requires the child to place a toy brick on a lever, which raises the lever to the top of the box, in which a toy becomes available. Only children who pass task 1 will go on to task 2. Noncompliance is scored from 1-6, and a higher score indicates greater non-compliance behaviors.
Change in anger behaviors of child as measured by the Tool task | Baseline, Post-test-2 (4 months after post test1)
  The parent and child complete two problem solving tasks that are graded in difficulty. The assessor explains the problem to the parent and gives the tool and apparatus to the child. The parent is instructed to allow the child to solve the problem independently, but provide as much help as they believe the child needs. Task 1 is the "tube task", in which the child has to insert a stick inside a tube to get a toy. Task 2 is the "clear box task" that requires the child to place a toy brick on a lever, which raises the lever to the top of the box, in which a toy becomes available. Only children who pass task 1 will go on to task 2. Anger is scored form 1-6, with a higher score indicating greater anger behaviors.
Change in anger/frustration behaviors specifically directed to parent as measured by the Tool task | Baseline, Post-test-2 (4 months after post test1)
  The parent and child complete two problem solving tasks that are graded in difficulty. The assessor explains the problem to the parent and gives the tool and apparatus to the child. The parent is instructed to allow the child to solve the problem independently, but provide as much help as they believe the child needs. Task 1 is the "tube task", in which the child has to insert a stick inside a tube to get a toy. Task 2 is the "clear box task" that requires the child to place a toy brick on a lever, which raises the lever to the top of the box, in which a toy becomes available. Only children who pass task 1 will go on to task 2. Anger/frustration behaviors specifically directed to parent is scored from 1-7, with a higher score indicating greater anger/frustration behaviors, .
Change in child coping as measured by the Tool task | Baseline, Post-test-2 (4 months after post test1)
  The parent and child complete two problem solving tasks that are graded in difficulty. The assessor explains the problem to the parent and gives the tool and apparatus to the child. The parent is instructed to allow the child to solve the problem independently, but provide as much help as they believe the child needs. Task 1 is the "tube task", in which the child has to insert a stick inside a tube to get a toy. Task 2 is the "clear box task" that requires the child to place a toy brick on a lever, which raises the lever to the top of the box, in which a toy becomes available. Only children who pass task 1 will go on to task 2. Coping is scored 1-5, with a higher score indicating greater coping behaviors.
Change in Child enthusiasm for the task as measured by the Tool task | Baseline, Post-test-2 (4 months after post test1)
  The parent and child complete two problem solving tasks that are graded in difficulty. The assessor explains the problem to the parent and gives the tool and apparatus to the child. The parent is instructed to allow the child to solve the problem independently, but provide as much help as they believe the child needs. Task 1 is the "tube task", in which the child has to insert a stick inside a tube to get a toy. Task 2 is the "clear box task" that requires the child to place a toy brick on a lever, which raises the lever to the top of the box, in which a toy becomes available. Only children who pass task 1 will go on to task 2. Enthusiasm is scored from 1-6, with a higher score indicating greater child enthusiasm for task.
Change in Child persistence behaviors related to attention as measured by the Tool task | Baseline, Post-test-2 (4 months after post test1)
  The parent and child complete two problem solving tasks that are graded in difficulty. The assessor explains the problem to the parent and gives the tool and apparatus to the child. The parent is instructed to allow the child to solve the problem independently, but provide as much help as they believe the child needs. Task 1 is the "tube task", in which the child has to insert a stick inside a tube to get a toy. Task 2 is the "clear box task" that requires the child to place a toy brick on a lever, which raises the lever to the top of the box, in which a toy becomes available. Only children who pass task 1 will go on to task 2. Persistence related to attention is scored from 1-5, with a higher score indicating greater child persistence behaviors related to attention.
Change in children's developing abilities in early language as assessed by the MacArthur-Bates Communicative Development Inventories (MB-CDIs) | Baseline, Post-test 2 (4 months after post test1)
  The MacArthur-Bates Communicative Development Inventories (MB-CDIs) are scored from 0 to 100 percentile, with a higher percentile indicating better language ability.
Change in Attention Disengagement to Positive and Negative Emotions as assessed by total time child looked at faces on screen during the looking task | Baseline, Post-test 2 (4 months after post test1)
  Children will complete a looking task in which fearful, happy, neutral, and control faces are presented individually on a screen. After the looking task, the child will complete an overlap task with the same stimuli. First, child's attention will be directed to the center of the screen with an 'attention-getter'. After attention is fixated for 1 second, a face appears centered on the screen. After 1 second, a distractor image appears in the periphery either to the right or left and remains on the screen for 3 seconds.
Change in Attention Disengagement to Positive and Negative Emotions as assessed by longest individual time child looked at faces on screen during the looking task | Baseline, Post-test 2 (4 months after post test1)
  Children will complete a looking task in which fearful, happy, neutral, and control faces are presented individually on a screen. After the looking task, the child will complete an overlap task with the same stimuli. First, child's attention will be directed to the center of the screen with an 'attention-getter'. After attention is fixated for 1 second, a face appears centered on the screen. After 1 second, a distractor image appears in the periphery either to the right or left and remains on the screen for 3 seconds.
Change in Attention Disengagement to Positive and Negative Emotions as assessed by the number of times child looked away from the faces and toward the distractor during the looking task | Baseline, Post-test 2 (4 months after post test1)
  Children will complete a looking task in which fearful, happy, neutral, and control faces are presented individually on a screen. After the looking task, the child will complete an overlap task with the same stimuli. First, child's attention will be directed to the center of the screen with an 'attention-getter'. After attention is fixated for 1 second, a face appears centered on the screen. After 1 second, a distractor image appears in the periphery either to the right or left and remains on the screen for 3 seconds.
Change in White matter structural integrity as indicated by fractional anisotropy measured by diffusion tensor imaging (DTI) magnetic resonance imaging (MRI) - uncinate fasciculus tract | Baseline, Post-test 2 (4 months after post test1)
  Anisotropy values range from 0 to 1, and a higher value indicates greater white matter structural integrity.
Change in White matter structural integrity as indicated by fractional anisotropy measured by diffusion tensor imaging (DTI) magnetic resonance imaging (MRI) - anterior thalamic radiation tract | Baseline, Post-test 2 (4 months after post test1)
  Anisotropy values range from 0 to 1, and a higher value indicates greater white matter structural integrity.
Change in White matter structural integrity as indicated by fractional anisotropy measured by diffusion tensor imaging (DTI) magnetic resonance imaging (MRI) - cingulum tract | Baseline, Post-test 2 (4 months after post test1)
  Anisotropy values range from 0 to 1, and a higher value indicates greater white matter structural integrity.
Change in White matter structural integrity as indicated by fractional anisotropy measured by diffusion tensor imaging (DTI) magnetic resonance imaging (MRI) - fornix tract | Baseline, Post-test 2 (4 months after post test1)
  Anisotropy values range from 0 to 1, and a higher value indicates greater white matter structural integrity.
Change in functional activity during rest as indicated by Resting Electroencephalography (EEG) value | Baseline, Post-test 2 (4 months after post test1)
  Following application of EEG caps and electrodes, resting EEG will be collected for 5 minute while an experimenter blows bubbles.
Change in functional activity when engaged in sustained activity as indicated by Event-related potential (ERP) negative central (NC) value recorded during EEG | Baseline, Post-test 2 (4 months after post test1)
  For ERP assessment, children view emotional faces in a passive viewing paradigm on a computer screen while EEG is performed.
Change in functional activity when engaged in sustained activity as indicated by Event-related potential (ERP) positive slow wave (PSW) value recorded during EEG | Baseline, Post-test 2 (4 months after post test1)
  For ERP assessment, children view emotional faces in a passive viewing paradigm on a computer screen while EEG is performed.

SECONDARY OUTCOMES:
Maternal depression as measured by the Beck's Depression Inventory | Post-test 1 (1-2 weeks post intervention)
  This 21-item multiple-choice self-report inventory. Total score ranges from 0-63 a higher number indicating greater depression.
Degree of chaos in the home as measured by the CHAOS questionnaire | Post-test 1 (1-2 weeks post intervention)
  The questionnaire includes 15 forced-choice items. Total score ranges from 15-90. A higher total score will indicate a home environment that is more chaotic
COVID-19 Exposure and Family Impact as assessed by the COVID-19 Exposure and Family Impact Survey - Exposure Score | Post-test 1 (1-2 weeks post intervention)
  This survey will measure family exposure to potentially traumatic aspects of COVID-19 and assesses the impact of the pandemic on the family. Parents will complete the survey. The Exposure Score ranges from 0 to 25, with a higher score indicating greater exposure.
COVID-19 Exposure and Family Impact as assessed by the COVID-19 Exposure and Family Impact Survey - Impact Score | Post-test 1 (1-2 weeks post intervention)
  This survey will measure family exposure to potentially traumatic aspects of COVID-19 and assesses the impact of the pandemic on the family. Parents will complete the survey. The Impact Score ranges from 12 to 60, with a higher score indicating greater impact.

CONTACTS AND LOCATIONS:
Overall Officials: Dana DeMaster, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No